CLINICAL TRIAL: NCT00803413
Title: Effect of Back School and Supervised Walking in Sedentary Women With Chronic Low Back Pain: a Randomized Controlled Trial.
Brief Title: Effect of Back School and Supervised Walking in Sedentary Women With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Mario Ferreira Junior, Hospital das Clínicas - São Paulo University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BSSW2002
Record Dates: First submitted 2008-11-07; First posted 2008-12-05 (Estimated); Results first posted 2008-12-05 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Back School; Walking; Physical activity
MeSH Terms: conditions — Motor Activity | interventions — Walking; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Back School (Other): Participants received weekly sessions of 45 minutes including: 15-minute lectures about basics of spine's anatomy, ergonomics, techniques of lifting and transportation of weights and volumes, body posture in several daily tasks and situations, and spine preventive care; 30 minutes of on-place supervised exercises for posture and spine flexibility (muscle stretching, relaxation, strengthening)
  Interventions: Behavioral: Back School Intervention
- Supervised Walking (Other): Participants received weekly sessions of 45 minutes including: 15-minute lectures about basics of physical activity, its advantages and benefits, barriers and facilitators, types and opportunities; 30 minutes of on-place supervised walking in group
  Interventions: Behavioral: Supervised Walking Intervention
- Back School and Walking (Other): Participants received weekly sessions of 90 minutes including: 30-minute lectures about basics of spine's anatomy, ergonomics, techniques of lifting and transportation of weights and volumes, body posture in several daily tasks and situations, spine preventive care, and about physical activity, its advantages and benefits, barriers and facilitators, types and opportunities; 30 minutes of on-place supervised exercises for posture and spine flexibility (muscle stretching, relaxation, strengthening); 30 minutes of on-place supervised walking in group
  Interventions: Behavioral: Back School and Walking
- Control Group (Other): Participants received weekly sessions of 45 minutes including lectures about: stress control, healthy nutrition (2 lectures), sleep hygiene and injury prevention; beside the 2-page folder content this group received no other information about LBP, BS or walking all along the follow-up.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Back School Intervention — Patients were submitted once a week for 5 consecutive weeks to sessions of 45 minutes including: 15-minute lectures about basics of spine's anatomy, ergonomics, techniques of lifting and transportation of weights and volumes, body posture in several daily tasks and situations, and spine preventive care; 30 minutes of on-place supervised exercises for posture and spine flexibility (muscle stretching, relaxation, strengthening)
  Other Names: BS
  Arms: Back School
Behavioral: Supervised Walking Intervention — Patients were submitted once a week for 5 consecutive weeks to sessions of 45 minutes including: 15-minute lectures about basics of physical activity, its advantages and benefits, barriers and facilitators, types and opportunities; 30 minutes of on-place supervised walking in group.
  Other Names: W
  Arms: Supervised Walking
Behavioral: Back School and Walking — Weekly sessions of 90 minutes including: 30-minute lectures about basics of spine's anatomy, ergonomics, techniques of lifting and transportation of weights and volumes, body posture in several daily tasks and situations, spine preventive care, and about physical activity, its advantages and benefits, barriers and facilitators, types and opportunities
  Other Names: BS+W
  Arms: Back School and Walking
Behavioral: Control Group — Weekly sessions of 45 minutes including lectures about: stress control, healthy nutrition (2 lectures), sleep hygiene and injury prevention.; beside the 2-page folder content this group received no other information about LBP, BS or walking all along the follow-up.
  Other Names: CG
  Arms: Control Group

SUMMARY:
Do Back School and/or supervised walking improve reported pain and spine flexibility in sedentary women with chronic low back pain (LBP)?

DETAILED DESCRIPTION:
From August 2002 to March 2004, one hundred nineteen volunteers sedentary women with chronic LBP and age ranging from 32 to 60 years old, randomly allocated to four groups of participants assigned as Back School (BS; N=28), Supervised Walking (W; N=32), Back School and Supervised Walking (BS+W; N=29), and Control Group (CG; N=30) were submitted to interventions once a week for 5 consecutive weeks and followed for up to 6 months. The groups BS, W, and BS+W received LBP-targeted lectures and on-place practical sessions of each respective intervention. CG received print information about LBP and 5 different lectures unrelated to LBP.

ELIGIBILITY:
Inclusion Criteria:

* Age range 30 to 60 years old
* LBP without any known organic cause for at least 3 months of duration
* Less than 90 minutes per week of regular physical activity of any intensity

Exclusion Criteria:

* Any known organic cause of LBP

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2002-08; Primary Completion 2003-06 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ferreira Junior, PhD, Principal Investigator — Hospital das Clínicas - São Paulo University School of Medicine
Locations (1):
- Center for Health Promotion - Hospital das Clínicas - FMUSP, São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2002 and March 2004, 351 women that attended 4 community centers located in the city of São Paulo, Brazil, responding to invitations by folders and voice announcements, filled a form with basic questions about physical activity and low back pain (LBP). After a clinical evaluation, 119 patients fulfilled the study criteria.
Groups:
- Backschool and Supervised Walking: Once a week for 5 consecitive weeks participants attended of 90 minutes including: 30-minute lectures about basics of spine's anatomy, ergonomics, techniques of lifting and transportation of weights and volumes, body posture in several daily tasks and situations, spine preventive care, and about physical activity, its advantages and benefits, barriers and facilitators, types and opportunities; 30 minutes of on-place supervised exercises for posture and spine flexibility (muscle stretching, relaxation, strengthening); 30 minutes of on-place supervised walking in group.
- Control Group: Once a week for 5 consecutive weeks participants attended sessions of 45 minutes including lectures about: stress control, healthy nutrition (2 lectures), sleep hygiene and injury prevention. This group also received a 2-page folder with print information about LBP prevention and control.
Period: Overall Period
Arm/Group | Back School | Supervised Walking | Backschool and Supervised Walking | Control Group
Started | 28 | 32 | 29 | 30
Completed | 28 | 32 | 29 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Back School | Supervised Walking | Backschool and Supervised Walking | Control Group | Total
Number analyzed (Participants) | 28 | 32 | 29 | 30 | 119
Age Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 32 | 30 | 119
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (7.3) | 47.2 (7.1) | 46.5 (7.5) | 46.8 (7.2) | 46.6 (7.4)
Gender [Number; unit: participants]
  Female | 28 | 29 | 32 | 30 | 119
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 28 | 29 | 32 | 30 | 119

OUTCOME MEASURES:

1. Secondary Outcome: Spine Flexibility (3rd Fingertip to Floor - 3FF).
Description: Patients in up-right position with joined feet and stretched out arms were asked to bend the spine as much as possible without bending the knees; the least achieved distance between the 3rd fingertip and the floor was measured in centimeters with a proper rule.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Back School | Supervised Walking | Backschool and Supervised Walking | Control Group
Number analyzed (Participants) | 28 | 32 | 29 | 30
centimeters | 20.8 (8.4) | 20.3 (8.1) | 20.4 (8.4) | 17.1 (13.0)

2. Primary Outcome: Intensity of Low Back Pain (LBP) Self-Estimated by Visual Analogical Scale (VAS)
Description: Patients were asked to indicate their perception about their LBP intensity with a cross on a line without marks, ranging from 1 (very light pain) through 10 (very strong pain)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Back School | Supervised Walking | Backschool and Supervised Walking | Control Group
Number analyzed (Participants) | 28 | 32 | 29 | 30
milimeters | 4.5 (3.3) | 4.2 (3.0) | 5.4 (2.7) | 3.9 (2.8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes